CLINICAL TRIAL: NCT04489472
Title: The Effect of a Dietary Supplement Rich in Nitric Oxide in Patients Diagnosed With Primary Ciliary Dyskinesia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Ricardo A. Mosquera, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-0382
Record Dates: First submitted 2020-07-02; First posted 2020-07-28 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Nitric oxide; Intranasal nitric oxide; Beet juice
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCD Group (Experimental)
  Interventions: Dietary Supplement: Beet-it Juice
- Control Group (Placebo Comparator)
  Interventions: Dietary Supplement: Beet-it Juice

INTERVENTIONS:
Dietary Supplement: Beet-it Juice — Patients will ingest 1 bottle (70ml) of beet-it juice (98% concentrated beet juice, 2% lemon juice containing 400 mg/6.5 mmol nitrate).

SUMMARY:
The purpose of this study is to determine the effect of a dietary supplement rich in nitric oxide (NO) on nasal nitric oxide and fractional exhaled nitric oxide (FeNO),on ciliary beat frequency assessed by high-speed digital video microscopy and on lung function assessed by spirometry in normal patients and patients with Primary ciliary dyskinesia (PCD).

ELIGIBILITY:
Inclusion Criteria:

Experimental group:

* PCD patients

Control Group:

* patients with no known chronic lung disease
* 18 years to 99 years

Exclusion Criteria(both PCD patients and control group):

* any other pulmonary co-morbidities and diseases entities like cystic fibrosis, nasal sinus surgery, nasal sinus hypoplasia/aplasia, deviated nasal septum, nasal polyps and with upper respiratory tract infection
* patients allergic to beet
* a known prolonged bleeding disorder.

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in nasal NO as measured by a chemiluminescence analyzer | Baseline,after beet juice consumption(1 hour after consumption)
Change in nasal NO as measured by a chemiluminescence analyzer | Baseline,after beet juice consumption( 2 hours after consumption)
Change in nasal FeNO as measured by using the NIOX MINO® Airway Inflammation Monitor | Baseline,after beet juice consumption(1 hour after consumption)
Change in nasal FeNO as measured by using the NIOX MINO® Airway Inflammation Monitor | Baseline,after beet juice consumption(2 hours after consumption)

SECONDARY OUTCOMES:
Change in ciliary beat frequency as measured using high-speed video-microscopy (HSVM) | after beet juice consumption(2 hours after consumption)
Change in lung function as measured by spirometry | Baseline,after beet juice consumption(2 hours after consumption)
  spirometry is used to assess how well your lungs work by measuring how much air you inhale,how much you exhale and how quickly you exhale

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Mosquera, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No